CLINICAL TRIAL: NCT04487301
Title: A Cross-Sectional Non-Interventional Study to Assess Walking Performance, Quality of Life, Vascular Function, and Lower Limb Arterial Calcification in Subjects With Peripheral Artery Disease and ESKD Receiving Hemodialysis
Brief Title: A Cross-Sectional Study to Assess Walking Performance in Subjects With Peripheral Artery and End Stage Kidney Disease
Status: Completed | Type: Observational
Sponsor: Sanifit Therapeutics S. A. (Other)
Responsible Party: Sponsor
Other Study IDs: SNFCT2020-07
Record Dates: First submitted 2020-07-20; First posted 2020-07-27 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Peripheral Artery Disease; End Stage Renal Disease on Dialysis
Keywords: PAD; Peripheral Artery Disease; End Stage Kidney Disease; End Stage Renal Disease; Dialysis
MeSH Terms: conditions — Peripheral Arterial Disease; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional, non-interventional study to assess walking performance, vascular function, and lower limb calcification in subjects with peripheral artery disease and end-stage kidney disease (PAD-ESKD) receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* ≥55 years of age or ≥45 years of age with diabetes
* Receiving maintenance HD in a clinical setting for at least 2 weeks prior to screening
* Resting ABI <0.90 in either leg OR Resting TBI <0.70 in either leg
* Symptomatic as characterized by a limitation in exercise performance

Exclusion Criteria:

* Above-ankle amputation
* Chronic limb-threatening ischemia (Rutherford 4-6)
* Non-ambulatory status
* A condition other than PAD that limits ability to walk
* Open or endovascular revascularization within 3 months prior to baseline.
* Illnesses, conditions, or planned surgeries within the study period that will interfere with the interpretation of the study results

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample of PAD-ESKD subjects
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-12 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk Test | Two six minute walk tests will be conducted separated by 5-7 days during Week 1 during the subject's participation of up to 4 weeks.
  Walking distance in meters completed over a duration of 6 minutes
Activity Patterns | Functional activity measurements will be collected daily beginning at the completion of screening and daily for the duration of the subject's participation of up to 4 weeks.
  Actigraphy measurements as 24 hour intervals of motion using an accelerometer device
Ankle Brachial Index | Will be conducted once in a vascular laboratory during the screening visit or visits during the subject's participation of up to 4 weeks
  Compares blood pressure in upper extremities and lower extremities
Toe Brachial Index | Will be conducted once in a vascular laboratory during the screening visit or visits during the subject's participation of up to 4 weeks
  Compares blood pressure in upper extremities and lower extremities
San Diego Claudication Questionnaire | Administered once during Day 1 of the screening visit during subject's participation of up to 4 weeks.
  Will categorize the subject's perception of the leg symptoms associated with PAD
Walking Impairment Questionnaire | Administered once during Week 1 during subject's participation of up to 4 weeks.
  Will evaluate the subjects personal perception of walking ability.
PAD Quality of Life | Administered once during Week 1 during subject's participation of up to 4 weeks.
  Will evaluate information about the subject's perception of social relationships, self-concepts and feelings, symptoms and limitations in physical functioning, fear and uncertainly, and positive adaptation.
EQ-SD-SL Health Questionnaire | Administered once during Week 1 during subject's participation of up to 4 weeks
  Will evaluate the subject's perception of overall health status, mobility, self-care, usual activities, pain or discomfort, and anxiety or depression.
Pulse Wave Velocity - Sub-Study | Will be conducted once in a vascular lab for subjects participating the in the sub-study during Week 3 of the subjects participation of 4 weeks.
  Measures arterial stiffness
Flow-Mediated Dilation - Sub-Study | Will be conducted once in a vascular lab for subjects participating the in sub-study during Week 3 of the subjects participation of 4 weeks.
  Measures the ability of blood vessels to dilate
Nitroglycerin-Medicated Dilation - Sub-Study | Will be conducted once in a vascular lab for subjects participating the in sub-study during Week 3 of the subjects participation of 4 weeks.
  Measures the ability of blood vessels to dilate after administration of nitroglycerin
Lower limb calcification measurements | Will be conducted once in subjects participating the in sub-study during Week 3 of the subjects participation of up to 4 weeks.
  A non-contrast computed tomography scan of the lower extremities will be evaluated for arterial calcification.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Gold, MD, Study Director — Sanifit Therapeutics
Locations (7):
- United States (7):
  - Valley Renal Medical Group, Northridge, California
  - Horizon Medical Research, Coral Gables, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - St Louis Kidney Care, St Louis, Missouri
  - Mountain Kidney & Hypertension Associates, Asheville, North Carolina
  - Houston Medical Research, Houston, Texas